CLINICAL TRIAL: NCT01224119
Title: A Multi-Center, Randomized, Pilot Study Evaluating Amplex Compared To Autograft Bone In Foot and Ankle Fusion Surgery
Brief Title: A Study Evaluating Amplex Compared To Autograft Bone In Foot and Ankle Fusion Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BioSurface Engineering Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMX-200
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Arthritis
Keywords: foot ankle arthritis bone graft
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amplex (synthetic bone graft) (Experimental)
  Interventions: Device: Amplex
- Autograft bone (Active Comparator)
  Interventions: Procedure: Autograft bone

INTERVENTIONS:
Device: Amplex — 225 micrograms of B2A per cc of ceramic granules
  Arms: Amplex (synthetic bone graft)
Procedure: Autograft bone — Bone is collected through a separate incision at the iliac crest or tibia.
  Arms: Autograft bone

SUMMARY:
The current research study evaluates an investigational medical device called Amplex B2A(TM) Peptide Enhanced Ceramic Granules ("Amplex") for use in foot and ankle fusion. Amplex is a synthetic bone graft material. The most frequently used graft material is bone collected from the patient (autograft). Autograft involves a secondary incision with the risks of infection and lasting pain.

The purpose of this study is to determine if Amplex is a safe and effective alternative to autograft.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for foot and ankle surgery described as either a single, double or triple arthrodesis of the ankle, subtalar, calcaneocuboid or talonavicular joints.
* Have the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol
* Have the ability to understand and provide written authorization for the use and disclosure of personal health information (PHI)
* Be a skeletally mature male or a non-pregnant, non-lactating female at least 18 years of age but not older than age 75
* If a woman is of childbearing potential (not amenorrheic for the previous 24 months or not surgically sterile), then she must:

  * Have a confirmed negative urine pregnancy test result prior to surgery and the administration of the study product
  * Agree to use a medically approved method of contraception for the duration of the initial follow-up period of the study
* Agree to participate in postoperative clinical and radiographic evaluations and comply with the required study regimen
* Have not been sufficiently responsive to an adequate trial of non-operative treatment (e.g. modified activity, analgesics, anti-inflammatories, bracing, orthotics, physiotherapy, vitamin supplements, or injections etc. prior to study enrollment).

Exclusion Criteria:

* Has a large bone deficit requiring a structural graft
* Charcot joints from neuropathic destruction.
* Previous fusion or osteotomy of the proposed site
* Requires osteotomy or fusion of the midfoot joints
* Morbidly obese (BMI >45 kg/m2)
* Women planning to become pregnant during the first year (12 months) following the procedure
* Female subjects of childbearing potential unwilling to use medically acceptable contraceptive methods (e.g., surgical sterilization, hormonal contraceptives, barrier methods, or intrauterine devices) so as to prevent pregnancy for 12 months following the study procedure
* Have at the time of surgery a systemic infection or local infection at the site of surgery
* Have an active history of systemic malignancy.
* Currently has untreated malignant neoplasm(s), or is currently undergoing radio- or chemotherapy or has been diagnosed with hypercalcemia.
* Have a medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study or potentially decrease survival or interfere with ambulation or rehabilitation (e.g., histories of transient ischemic attack, stroke or liver disease)
* Has a known complication of diabetes (e.g. retinopathy, renal failure, neuropathic complication in lower limb).
* Uncontrolled diabetes. If the patient has been diagnosed with diabetes, they must have an Hgb A1C level less than 7 to participate.
* Have a known hypersensitivity to any of the components of the product [e.g., Hydroxyapatite (HA): Tricalcium Phosphate (TCP) ceramic granule] or a known titanium allergy
* Receiving active treatment with a drug known to interfere with bone metabolism (e.g. long-term steroid therapy, methotrexate).
* Have a history of any severe allergy or anaphylaxis, or a history of hypersensitivity to protein pharmaceuticals (e.g., monoclonal antibodies or gamma globulins, recombinant BMPs)
* Being treated with a bone growth stimulator
* Have a medical condition requiring radiation, chemotherapy or immunosuppression.
* Have obvious and/or documented alcohol or illicit drug addictions
* Are prisoners
* Have participated in clinical studies evaluating investigational devices, pharmaceuticals or biologics within 3 months of enrollment
* Have previously been treated with, or exposed to, therapeutic levels of Bone Morphogenetic Proteins (BMPs), i.e., synthetic or recombinant
* Have a documented medical history of or radiographic evidence of a metabolic bone disease (e.g., avascular necrosis, osteoporosis or osteopenia) or other condition that would negatively impact the bone healing process (e.g. history of Paget's disease, osteomalacia, or other osteodystrophy) or preclude the subject from receiving screw fixation.
* Require chronic SQ or IV heparin therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Radiographic fusion | 6 months
  An independent radiologist will assess radiographic fusion based upon CT imaging.
Ankle Osteoarthritis Questionnaire | 6 months
  This is a questionnaire completed by the subject. It consists of a number of questions concerning the amount of pain in the foot and its effect on functional activities.

SECONDARY OUTCOMES:
Ankle Osteoarthritis Questionnaire | 12 months
  The is a questionnaire completed by the subject. Its asks a series of questions about pain and function of the treated foot or ankle.
Radiographic fusion | 9-12 months
  Radiographic fusion will be assess by a blinded indpenendent radiologists, using CT and X-ray images. The investigator will also assess fusion based on the images and also the overall condition of the subject.
Various blood tests | PreOp through 6 months
  Small amounts of blood will be collected at study visits to identify possible changes in blood chemistry, liver function and antibody formation.

CONTACTS AND LOCATIONS:
Overall Officials: David M Hooper, PhD, Study Director — BioSurface Engineering Technologies, Inc; Mark Glazebrook, MD, Principal Investigator — Queen Elizabeth II Health Sciences Center Halifax Infirmary
Locations (1):
- Dr. Mark Glazebrook, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Glazebrook M, Younger A, Wing K, Lalonde KA. A prospective pilot study of B2A-coated ceramic granules (Amplex) compared to autograft for ankle and hindfoot arthrodesis. Foot Ankle Int. 2013 Aug;34(8):1055-63. doi: 10.1177/1071100713481459. Epub 2013 Mar 5. PMID 23463779